CLINICAL TRIAL: NCT03347084
Title: Study of Non-Invasive Deep Brain Stimulation with Low Intensity Focused Ultrasound Pulse (LIFUP) for Mild Cognitive Impairment (MCI) and Mild Alzheimer's Disease (AD)
Brief Title: Deep Brain Stimulation with LIFUP for Mild Cognitive Impairment and Mild Alzheimer's Disease
Acronym: LIFUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Taylor Kuhn, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 16-001314
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Brain Imaging; Mild Cognitive Impairment; Alzheimer Disease; Deep Brain Stimulation
Keywords: DBS; brain imaging; Memory; fMRI
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Microscopy, Fluorescence, Multiphoton

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two LIFUP pulsing paradigms: one that excites the activity of hippocampal neurons ("Paradigm A"), or a second that inhibits them ("Paradigm B"). The participants will then be administered four successive LIFUP treatments while the participants are in a functional magnetic resonance imaging (MRI).
Who Masked: Participant
Masking Description: Participants and the participants' caregivers will be blinded to arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Excitation (Active Comparator): Excitation Paradigm: LIFUP excites the activity of hippocampal neurons.
  Interventions: Device: Excitation
- Inhibition (Active Comparator): Inhibition Paradigm: LIFUP inhibits the activity of hippocampal neurons.
  Interventions: Device: Inhibition

INTERVENTIONS:
Device: Excitation — Administration of LIFUP, a method of deep brain stimulation, according to excitation paradigms using the following parameters: Tone Burst Duration = 50ms; Pulse Repetition Frequency = 10Hz; ISPTA = 720 mW/cm2. Four treatments of thirty seconds each, with two-minute intervals between treatment (20 minutes, approximately)
  Other Names: Low Intensity Focused Ultrasound Pulse
  Arms: Excitation
Device: Inhibition — Administration of LIFUP, a method of deep brain stimulation, according to inhibition paradigms using the following parameters: Tone Burst Duration = 50ms and Pulse Repetition Frequency = 10Hz. Four treatments of thirty seconds each, with two-minute intervals between treatment (20 minutes, approximately)
  Other Names: Low Intensity Focused Ultrasound Pulse
  Arms: Inhibition

SUMMARY:
The purpose of the proposed study is to determine the feasibility of brief brain stimulation, using a device called Low Intensity Focused Ultrasound Pulsation (LIFUP), for persons with mild cognitive impairment (MCI) or mild (early-stage) Alzheimer's disease (AD). As a secondary aim, the investigators will explore whether this brief intervention is associated with improvements in cognitive functioning immediately and one week following the intervention.

Subjects will be randomly assigned to one of two experimental groups: either the LIFUP administration will be designed to increase the activity of neurons in a certain part of the brain or decrease the activity of neurons.

The investigators will study up to 8 subjects with MCI or mild AD. Initially, subjects will undergo a screening assessment with a study physician to determine medical and psychiatric history, establish AD diagnosis, and undergo a blood draw, if standard recent labs for dementia and EKG are unavailable. Subjects that meet criteria and agree to participate in the study will undergo a follow-up visit. In the baseline measurement visit, participants will first undergo neuropsychological testing. Participants will be randomly assigned to one of two LIFUP pulsing paradigms. Participants will then be administered four successive LIFUP treatments while the participants are in a functional magnetic resonance imaging (MRI). Sixty minutes following the administration, participants will undergo a second neuropsychological test. A final follow-up assessment will be administered at one week.

DETAILED DESCRIPTION:
Alzheimer disease (AD) is a neurodegenerative condition and the most common cause of dementia or a functional impairment in memory and other cognitive abilities. Prior to developing the functional impairment of dementia, patients develop mild cognitive impairment (MCI), which increases the risk for developing the functional impairment of dementia. Deep brain stimulation (DBS) is of interest as a potential therapeutic option for MCI and AD because it can directly target and modulate the activity of brain structures implicated in memory functioning.

Recently there have been multiple reports that DBS of different locations within the brain may be effective in improving symptoms characteristic of dementia (e.g., Heschman et al., 2013). For example, Laxton et al. (2010) performed DBS in the fornix/hypothalamus of six persons with AD in a phase I clinical trial. The investigators hypothesized that stimulation of the fornix would alter the activity of the medial temporal memory circuits, and thus delay and/or reverse memory loss. After 6-12 months, the investigators noted improvement or slowing in the progression of AD in some of the research participants, as measured by two commonly-used assessments of global cognitive function. In a recent literature review, Laxton et al. (2013) also described several additional studies demonstrating that DBS of the fornix or nucleus of Meynert or subthalamic nucleus influences the pathologic neurological circuits involved in AD.

Four separate groups recently have published reports concluding that ultrasound improves amyloid-β clearance in mouse models and restores memory (e.g., Leinenga & Götz, 2015). This finding raises the question of whether one method of DBS, Low Intensity Focused Ultrasound Pulse (LIFUP), could improve cognition in patients with AD, which is characterized by abnormal deposition of amyloid plaques in brain regions controlling memory and thinking. The use of LIFUP in animal models is well described (Bystritsky et al., 2014). LIFUP is able to penetrate the human skull and reach deep structures within the temporal therapeutic window. The structures that are reachable by LIFUP include the temporal cortices, hippocampus, thalamus, and subthalamic nuclei, all of which are implicated in the pathophysiology of AD. The Food and Drug Administration (FDA) recently approved an investigational device exemption (IDE) to begin a feasibility and safety trial of LIFUP for persons with refractory seizures.

Although symptomatic treatments are available for AD, their modest effects are temporary and there is a need for more effective interventions. In the current project, the investigators propose to use the FDA-approved protocol to:

1. Determine the feasibility of a brief LIFUP intervention (four stimulations of 30 seconds each, with 2-minute intervals between each treatment) for persons with MCI or mild (early-stage) AD.
2. As a secondary aim, the investigators will explore whether this brief LIFUP intervention is associated with improvements on neuropsychological measures of cognitive functioning immediately following the intervention.

To investigate these aims, subjects with MCI or mild AD will be enrolled. Subjects will be randomized using a single-blind design, to one of two LIFUP pulsing paradigms in which activity of neurons in a certain part of the brain are either increased. Subjects will then be administered four successive LIFUP treatments while the subjects are in a functional magnetic resonance imaging (MRI). Neuropsychological assessments will be performed at baseline, immediately after LIFUP is administered, and one week following the conclusion of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment or mild (early-stage) AD diagnosis through medical record review
* Agreement to participate in a clinical and brain imaging study.
* Age 55 years or older.
* No significant cerebrovascular disease as determined by a modified Ischemic Score of ≤ 4.
* Availability of a study partner (next of kin, family member) to attend all visits and to provide surrogate consent should it be determined that the participant does not have capacity.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Screening laboratory tests and ECG without significant abnormalities that might interfere with the study.
* Use of cholinesterase inhibitors for AD (Aricept, Namenda, etc.) will be allowed as long as the participant has been on a stable dose for at least two months.
* There must be a family member or caregiver available to make sure the participant gives informed consent, and in case the participant develops cognitive impairment that interferes with independent study participation.

Exclusion Criteria:

* Evidence of any other major neurologic or other physical illness that could produce cognitive deterioration, except for mild cognitive impairment (MCI) and any history of stroke or diabetes.
* History of myocardial infarction within the previous year or unstable cardiac disease.
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100), history of significant liver disease, clinically significant pulmonary disease, diabetes, or cancer.
* Major psychiatric disorders, such as bipolar disorder or schizophrenia, or persons with current untreated major depression
* Current diagnosis or significant history of alcoholism or drug dependence.
* Participants taking medications known to influence cognitive functioning will be excluded. Medications that will be excluded include: centrally active beta-blockers, narcotics, clonidine, anti-Parkinsonian medications, benzodiazepines, systemic corticosteroids, and medications with significant anticholinergic effects, anti-convulsants, or warfarin. During the screening visit, physicians will review all medications and determine whether the type, dose, and interaction of medications are likely to impact cognition and determine exclusion based on these factors.
* Use of any investigational drugs within the previous month or longer, depending on the drug's half-life.
* Contraindication for fMRI scan (e.g. metal in body, claustrophobia).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fMRI brain scan to 40 minutes. | 40 Minutes
  Functional MRI of the brain will be obtained throughout the LIFUP session for the purposes of image acquisition.

SECONDARY OUTCOMES:
Change from baseline in Hopkins Verbal Learning Test-Revised45 (HVLT-R) | 60 Minutes, 1 Week
  The Hopkins Verbal Learning Test-Revised will provide a measure of verbal memory. It requires recall of a series of 12 words over three learning trials, free recall after a 25-minute delay, and a recognition trial. There are 6 equivalent alternate forms.
Change from baseline in Brief Visual Memory Test-Revised | 60 Minutes, 1 Week
  The Brief Visual Memory Test-Revised will provide a measure of visual memory. In three learning trials, the respondent views 6 geometric figures for 10 seconds and is asked to draw as many of the figures as possible from memory in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Last, a Recognition Trial, in which the respondent is asked to identify which of 12 figures were included among the original geometric figures, is administered. There are 6 equivalent alternate forms.
Change from baseline in Geriatric Anxiety Inventory (GAI) | 60 Minutes, 1 Week
  Geriatric Anxiety Inventory (GAI) will be used as a measure to ensure that pre-LIFUP/pre-MRI anxiety is not significantly impacting performance on the first neuropsychological assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Taylor P Kuhn, PhD, Principal Investigator — UCLA Longevity Center
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization (WHO). Dementia cases set to triple by 2050 but still largely ignored. Geneva, Switzerland; 2012.
- [Background] Prince M, Bryce R, Ferri C. World Alzheimer report. Alzheimer's Disease International; 2011 Sep.
- [Background] Okun MS. Deep-brain stimulation for Parkinson's disease. N Engl J Med. 2013 Jan 31;368(5):483-4. doi: 10.1056/NEJMc1214078. No abstract available. PMID 23363512
- [Background] Halpern C, Hurtig H, Jaggi J, Grossman M, Won M, Baltuch G. Deep brain stimulation in neurologic disorders. Parkinsonism Relat Disord. 2007 Feb;13(1):1-16. doi: 10.1016/j.parkreldis.2006.03.001. Epub 2006 Dec 1. PMID 17141550
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Greenberg BD, Malone DA, Friehs GM, Rezai AR, Kubu CS, Malloy PF, Salloway SP, Okun MS, Goodman WK, Rasmussen SA. Three-year outcomes in deep brain stimulation for highly resistant obsessive-compulsive disorder. Neuropsychopharmacology. 2006 Nov;31(11):2384-93. doi: 10.1038/sj.npp.1301165. Epub 2006 Jul 19. PMID 16855529
- [Background] Stephen JH, Halpern CH, Barrios CJ, Balmuri U, Pisapia JM, Wolf JA, Kampman KM, Baltuch GH, Caplan AL, Stein SC. Deep brain stimulation compared with methadone maintenance for the treatment of heroin dependence: a threshold and cost-effectiveness analysis. Addiction. 2012 Mar;107(3):624-34. doi: 10.1111/j.1360-0443.2011.03656.x. PMID 21919988
- [Background] Pisapia JM, Halpern CH, Williams NN, Wadden TA, Baltuch GH, Stein SC. Deep brain stimulation compared with bariatric surgery for the treatment of morbid obesity: a decision analysis study. Neurosurg Focus. 2010 Aug;29(2):E15. doi: 10.3171/2010.5.FOCUS10109. PMID 20672917
- [Background] Hescham S, Lim LW, Jahanshahi A, Blokland A, Temel Y. Deep brain stimulation in dementia-related disorders. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2666-75. doi: 10.1016/j.neubiorev.2013.09.002. Epub 2013 Sep 20. PMID 24060532
- [Background] Hardenacke K, Kuhn J, Lenartz D, Maarouf M, Mai JK, Bartsch C, Freund HJ, Sturm V. Stimulate or degenerate: deep brain stimulation of the nucleus basalis Meynert in Alzheimer dementia. World Neurosurg. 2013 Sep-Oct;80(3-4):S27.e35-43. doi: 10.1016/j.wneu.2012.12.005. Epub 2012 Dec 12. PMID 23246738
- [Background] Fontaine D, Deudon A, Lemaire JJ, Razzouk M, Viau P, Darcourt J, Robert P. Symptomatic treatment of memory decline in Alzheimer's disease by deep brain stimulation: a feasibility study. J Alzheimers Dis. 2013;34(1):315-23. doi: 10.3233/JAD-121579. PMID 23168448
- [Background] Sankar T, Tierney TS, Hamani C. Novel applications of deep brain stimulation. Surg Neurol Int. 2012;3(Suppl 1):S26-33. doi: 10.4103/2152-7806.91607. Epub 2012 Jan 14. PMID 22826807
- [Background] Laxton AW, Lozano AM. Deep brain stimulation for the treatment of Alzheimer disease and dementias. World Neurosurg. 2013 Sep-Oct;80(3-4):S28.e1-8. doi: 10.1016/j.wneu.2012.06.028. Epub 2012 Jun 19. PMID 22722036
- [Background] Vitek JL. Long-term benefit from deep brain stimulation of the subthalamic nucleus: is it for everyone? Alzheimers Res Ther. 2012 May 9;4(3):13. doi: 10.1186/alzrt111. PMID 22574875
- [Background] Smith GS, Laxton AW, Tang-Wai DF, McAndrews MP, Diaconescu AO, Workman CI, Lozano AM. Increased cerebral metabolism after 1 year of deep brain stimulation in Alzheimer disease. Arch Neurol. 2012 Sep;69(9):1141-8. doi: 10.1001/archneurol.2012.590. PMID 22566505
- [Background] Lyons MK. Deep brain stimulation: current and future clinical applications. Mayo Clin Proc. 2011 Jul;86(7):662-72. doi: 10.4065/mcp.2011.0045. Epub 2011 Jun 6. PMID 21646303
- [Background] Laxton AW, Tang-Wai DF, McAndrews MP, Zumsteg D, Wennberg R, Keren R, Wherrett J, Naglie G, Hamani C, Smith GS, Lozano AM. A phase I trial of deep brain stimulation of memory circuits in Alzheimer's disease. Ann Neurol. 2010 Oct;68(4):521-34. doi: 10.1002/ana.22089. PMID 20687206
- [Background] Laxton AW, Lipsman N, Lozano AM. Deep brain stimulation for cognitive disorders. Handb Clin Neurol. 2013;116:307-11. doi: 10.1016/B978-0-444-53497-2.00025-5. PMID 24112904
- [Background] Leinenga G, Gotz J. Scanning ultrasound removes amyloid-beta and restores memory in an Alzheimer's disease mouse model. Sci Transl Med. 2015 Mar 11;7(278):278ra33. doi: 10.1126/scitranslmed.aaa2512. PMID 25761889
- [Background] Wood H. Alzheimer disease: scanning ultrasound elicits amyloid-beta clearance in mice. Nat Rev Neurol. 2015 May;11(5):247. doi: 10.1038/nrneurol.2015.54. Epub 2015 Mar 31. No abstract available. PMID 25825222
- [Background] Lin WT, Chen RC, Lu WW, Liu SH, Yang FY. Protective effects of low-intensity pulsed ultrasound on aluminum-induced cerebral damage in Alzheimer's disease rat model. Sci Rep. 2015 Apr 15;5:9671. doi: 10.1038/srep09671. PMID 25873429
- [Background] Burgess A, Dubey S, Yeung S, Hough O, Eterman N, Aubert I, Hynynen K. Alzheimer disease in a mouse model: MR imaging-guided focused ultrasound targeted to the hippocampus opens the blood-brain barrier and improves pathologic abnormalities and behavior. Radiology. 2014 Dec;273(3):736-45. doi: 10.1148/radiol.14140245. Epub 2014 Sep 15. PMID 25222068
- [Background] Bystritsky A, Korb AS, Douglas PK, Cohen MS, Melega WP, Mulgaonkar AP, DeSalles A, Min BK, Yoo SS. A review of low-intensity focused ultrasound pulsation. Brain Stimul. 2011 Jul;4(3):125-36. doi: 10.1016/j.brs.2011.03.007. Epub 2011 Apr 1. PMID 21777872
- [Background] Rosen WG. Verbal fluency in aging and dementia. J Clin Neuropsychol. 1980;2(2):135-46. doi: 10.1080/01688638008403788.
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed). Washington, DC: American Psychiatric Association; 2013.
- [Background] Small GW, Rabins PV, Barry PP, Buckholtz NS, DeKosky ST, Ferris SH, Finkel SI, Gwyther LP, Khachaturian ZS, Lebowitz BD, McRae TD, Morris JC, Oakley F, Schneider LS, Streim JE, Sunderland T, Teri LA, Tune LE. Diagnosis and treatment of Alzheimer disease and related disorders. Consensus statement of the American Association for Geriatric Psychiatry, the Alzheimer's Association, and the American Geriatrics Society. JAMA. 1997 Oct 22-29;278(16):1363-71. PMID 9343469
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Bushberg JT, Seibert JA, Leidholdt EM Jr., Boone JM. The essential physics of medical imaging (3rd ed). Philadelphia, PA: Lippincott Williams & Wilkins; 2012.
- [Background] American Institute of Ultrasound in Medicine. Official statement on "Safety in training and research." http://www.aium.org/officialStatements/36. Published 2012 Apr 1; Accessed 2015 Sep 22.
- [Background] Yoo SS, Bystritsky A, Lee JH, Zhang Y, Fischer K, Min BK, McDannold NJ, Pascual-Leone A, Jolesz FA. Focused ultrasound modulates region-specific brain activity. Neuroimage. 2011 Jun 1;56(3):1267-75. doi: 10.1016/j.neuroimage.2011.02.058. Epub 2011 Feb 24. PMID 21354315
- [Background] Korb AS, Shellock FG, Cohen MS, Bystritsky A. Low-intensity focused ultrasound pulsation device used during magnetic resonance imaging: evaluation of magnetic resonance imaging-related heating at 3 Tesla/128 MHz. Neuromodulation. 2014 Apr;17(3):236-41; discussion 241. doi: 10.1111/ner.12075. Epub 2013 May 10. PMID 23663228
- [Background] Zeineh MM, Engel SA, Thompson PM, Bookheimer SY. Unfolding the human hippocampus with high resolution structural and functional MRI. Anat Rec. 2001 Apr;265(2):111-20. doi: 10.1002/ar.1061. PMID 11323773
- [Background] Ekstrom A. How and when the fMRI BOLD signal relates to underlying neural activity: the danger in dissociation. Brain Res Rev. 2010 Mar;62(2):233-44. doi: 10.1016/j.brainresrev.2009.12.004. Epub 2009 Dec 21. PMID 20026191
- [Background] Greicius MD, Srivastava G, Reiss AL, Menon V. Default-mode network activity distinguishes Alzheimer's disease from healthy aging: evidence from functional MRI. Proc Natl Acad Sci U S A. 2004 Mar 30;101(13):4637-42. doi: 10.1073/pnas.0308627101. Epub 2004 Mar 15. PMID 15070770
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396
- [Background] Murphy K, Birn RM, Handwerker DA, Jones TB, Bandettini PA. The impact of global signal regression on resting state correlations: are anti-correlated networks introduced? Neuroimage. 2009 Feb 1;44(3):893-905. doi: 10.1016/j.neuroimage.2008.09.036. Epub 2008 Oct 11. PMID 18976716
- [Background] Brandt J, Benedict R. Hopkins Verbal Learning Test-Revised: Professional Manual. PAR: Florida; 2001.
- [Background] 46Benedict RHB. Brief Visuospatial Memory Test - Revised: Professional Manual. Lutz, FL: Psychological Assessment Resources, Inc; 1997
- [Background] Pachana NA, Byrne GJ, Siddle H, Koloski N, Harley E, Arnold E. Development and validation of the Geriatric Anxiety Inventory. Int Psychogeriatr. 2007 Feb;19(1):103-14. doi: 10.1017/S1041610206003504. PMID 16805925
- See also: Analysis Group, Oxford, UK. FMRIB Software Library v5.0. — http://fsl.fmrib.ox.ac.uk/fsl/fslwiki/